### **INCREASED HEALTH AND SAFETY DURING COVID-19**

#### Remote Assessment

- You will receive the wearable or package via post or courier
- Please leave the package for 72 hours before opening
- All devices will be sanitized before being sent (person sending wearing PPE)

### **Lab Based testing only**

- All research will adhere to local (university) and national (government) guidance
- We will require you to confirm you have had no: contact with anyone testing positive or have/had symptoms of COVID-19 in the previous 14 days.
- All participants and researchers will be required to wear a facemask at all times. (Researchers will be wearing appropriate PPE)
- The laboratory including **all equipment will be cleaned** before and after each participant, with **extra time** given to ensure health and safety maintained and **no mixing between participants**.
- We will maintain social distancing at all times (1 meter plus).
- You may withdraw at any time without reason

If you need help or are worried about the virus, we can provide signposting to the appropriate services within the university - ask4help@northumbria.ac.uk

https://www.northumbria.ac.uk/study-at-northumbria/support-for-students/counselling-and-mental-health-support/self-help-students/counselling-and-mental-health-support/self-help-students/counselling-and-mental-health-support/self-help-students/counselling-and-mental-health-support/self-help-students/counselling-and-mental-health-support/self-help-students/counselling-and-mental-health-support/self-help-students/counselling-and-mental-health-support/self-help-students/counselling-and-mental-health-support/self-help-students/counselling-and-mental-health-support/self-help-students/counselling-and-mental-health-support-self-help-students/counselling-and-mental-health-support-self-help-students/self-help-stude

Computer and Information Science Northumbria University Newcastle upon Tyne

NEI 8ST

Telephone: 0191 227 3642

## **PARTICIPANT CONSENT FORM**

# THE USE OF WEARABLES AS OBJECTIVE TOOLS IN MONITORING OF SPORTS RELATED CONCUSSION

Name of researcher taking consent:

We are asking you to take part in a technology-based concussion related study as part of a PhD project.

Please be sure you have read the accompanying information sheet, it explains why we are doing this research and what we are asking you to do. If you find reading or understanding the information difficult, please ask a family member or friend to read it to you.

Please feel free to ask the research team any questions.

Remember, there is no obligation for you to take part in this research study. You are free to remove yourself from the study at any time.

Name of PhD Student: Dylan Powell Email: <a href="mailto:d.powell@northumbria.ac.uk">d.powell@northumbria.ac.uk</a> Name of Supervisor: Alan Godfrey

Email: alan.godfrey@northumbria.ac.uk

Title of Project: The Use of Wearables as Objective Tools in Monitoring of Sports Related Concussion

| | Initial | |
|---|---|---|
| Please initial the boxes that apply to you | Consent | Decline |
| I confirm that I have read and understand the information sheet dated | | |
| (version) for the above study. I have had the opportunity to consider the | | |
| information, ask questions and have had these answered satisfactorily and confirm that | | |
| I have not had contact with anyone testing positive or have/had symptoms of COVID- | | |
| 19 in the previous 14 days. | | |
| I understand that my participation is voluntary and that I am free to withdraw at any | | |
| time without giving any reason, without my medical care or legal rights being affected. | | |
| In the event that a <b>new potential medical problem</b> is found as a result of my | | |
| participation in this study I agree that the research team may inform my GP or relevant | | |
| medical professional about this. | | |
| I understand that individuals from this study research team at Northumbria University | | |
| may look at my data collected during the study. | | |
| I agree to have appropriate sections of the Balance Assessment procedures videoed for | | |
| verification purposes. | | |
| I agree to anonymous movement data to be taken during my involvement within the | | |
| study named above which may be during a match or another university setting | | |
| (including club) or my habitual environment, e.g. my home. | | |
| I agree to participate in this study. | | |
| ADDITIONAL (OPTIONAL) STUDIES | | |
| I understand it will not be possible to connect my name to data taken for any future | | |
| analysis for additional studies/work after it has been taken. | | |
| Any additional study may make use of the anonymous data collected from your | | |
| involvement in this current study, i.e. your activity data from the activity monitors, your | | |
| gender, age, weight, etc. These are classified as secondary analysis studies i.e. examining | | |
| the data in different ways. This is done so anonymously, and you will not be contacted | | |
| for any further information. All data is stored for 10 years after which it is disposed of if | | |
| not regularly used. | | |

| Participant: |
|------------------------|
| Signed |
| Printed name |
| Date |
| Person taking consent: |
| Printed name |
| Signed |
| Date |
| Designation |